CLINICAL TRIAL: NCT04630119
Title: Prospective Analysis of Pre-treatment Quality of Life, Presenteeism, and Emotional Health Due to Chronic Neck Pain in Homemakers- An Indian Tertiary Care Hospital Perspective
Brief Title: Prospective Analysis of Quality of Life, Presenteeism, and Emotional Health Due to Chronic Neck Pain in Homemakers
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health and Neuro Sciences, India (Other)
Responsible Party: Principal Investigator, Dhritiman Chakrabarti, Assistant Professor, National Institute of Mental Health and Neuro Sciences, India
Other Study IDs: AIIMSRPR/IEC/2019/327
Record Dates: First submitted 2020-11-09; First posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Chronic Neck Pain
Keywords: chronic neck pain,; homemakers; presenteeism; quality of life
MeSH Terms: interventions — Mental Health; Presenteeism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group of female homemakers with chronic neck pain: All female patients aged between 18-55 years with chronic neck pain (pain lasting for more than 3months) who were homemakers were included in the study. All participants reported the presence of pain in the preceding one week
  Interventions: Other: Questionnaires on quality of life, emotional health and presenteeism

INTERVENTIONS:
Other: Questionnaires on quality of life, emotional health and presenteeism — After obtaining informed consent, a pro forma consisting of the socio-demographic details and pre-treatment assessment questionnaire (including Visual analog scale The Medical Outcomes Study Short-Form Health Survey The hospital anxiety and depression scale Work functioning impairment scale) was filled for each subject.

SUMMARY:
Chronic pain is defined as persistent or recurrent pain lasting longer than 3 months as per ICD11 and includes seven categories of pain. Chronic musculoskeletal pain is one of them. Neck pain is one of the top five causes of chronic pain yet few clinical trials are dedicated solely to neck pain. Chronic neck pain not only leads to neuromuscular dysfunction but also psychological distress and fear-avoidance all contributing to reduced quality of life, emotional health, and productivity of a person. Absenteeism and presenteeism are both measures of work productivity of a person but presenteeism is more significant where being absent from work is not a feasible option like in the case of homemakers.

Homemakers are often neglected but they constitute an essential part of society. Although they do not have a formal occupation, they perform a multitude of ergonomically stressful activities leading to different types of musculoskeletal pain. Being mostly a silent sufferer, they often seek medical help when the pain becomes chronic and affects different areas of health thereby necessitating a holistic management approach.

In the Central Indian cultural scenario, a homemaker rarely takes complete rest from her household chores. So presenteeism can be used as a marker for work productivity. This study aims to analyze the impact of chronic neck pain in the pre-treatment quality of life, presenteeism, and emotional health in homemakers and to find the association of the findings with the cause and severity of chronic neck pain.

DETAILED DESCRIPTION:
Chronic pain is defined as a persistent or recurrent pain lasting longer than 3 months as per ICD11 and constitutes of seven categories of pain including musculoskeletal pain. Neck pain is one of the top five causes of chronic pain which globally affects 332 million and ranks 4-6th as a cause of Years Lived with Disability. It has been described by the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders as 'pain located in the anatomical region of the neck with or without radiation to the head, trunk, and upper limbs. Chronic neck pain not only leads to neuromuscular dysfunction but also psychological distress and fear-avoidance all contributing to reduced quality of life and emotional health.

Chronic pain expectedly affects the work productivity of an individual. Work productivity is measured by either 'absenteeism' or 'presenteeism'. Absenteeism (absence from work) is calculated by missed days at work and presenteeism means being present at work while experiencing health complaints or to put it simply 'not unwell enough" to skip work when sick. Presenteeism is commonly interpreted through various scales of pain, cognition, and quality of life. The highest rate of presenteeism across various sectors has been reported in human service organizations that deal with care, welfare, and education. The last decade has seen a surge in interest in presenteeism and the concept has received both positive and negative criticism. High presenteeism ensures excellent attendance at work but also signifies a higher workload and poor work-life balance along with variations in personal work ethics. Presenteeism has been variously studied across different disease conditions and specific ergonomic populations but there are very limited studies on homemakers.

Homemakers along with students and retirees are considered a part of the Out of the labor force (OLF) of the society who do not have an income and are hence formally unemployed. However, in a patriarchal society like India, women homemakers often perform a multitude of roles (parental, caretaker, household) which are comparable to that of paid domestic help and can be classified as an occupation on its own. Observing from an ergonomic point of view, homemakers engage in activities that involve prolonged awkward postures as well as repetitive movements which are risk factors for various musculoskeletal pain of the neck, back, and limbs. But unlike other professions, there is no externally imposed time frame or formal 'breaks' which prevents a homemaker from taking a leave. Thus despite the biomechanical and psychosocial stress, homemakers continue their chores and seek help only when the pain is chronic and unbearable. So presenteeism instead of absenteeism is a more appropriate and reliable marker for work productivity amongst homemakers.

Although there are studies to see the prevalence of neck pain in the world, there are few clinical studies dedicated solely to neck pain especially in a specific population of homemakers more so in Central India.

The aim of this study was to analyse the impact of chronic neck pain in the pre-treatment quality of life, presenteesism and emotional health in homemakers and to find the association of the findings with the cause and severity of chronic neck pain.

All patients who met the inclusion criteria were approached with the study. After obtaining informed consent, a pro forma consisting of the socio-demographic details and pre-treatment assessment questionnaire (including Visual analog scale The Medical Outcomes Study Short-Form Health Survey The hospital anxiety and depression scale Work functioning impairment scale) was filled for each subject. The record was maintained based on a serial number given to each patient. Routine blood investigations (complete blood count, fasting blood sugar, renal, liver, and thyroid function test was done for all. X-ray of the cervical spine (AP and Lateral views) was prescribed. The final diagnosis was noted in subsequent follow-ups at OPD .

The results were then co related with the cause of chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

Patients of chronic neck pain (pain more than 3 months) Pain present in the last one week. Female gender. Homemakers Age between18-55 years

Exclusion Criteria:

Pregnant. Uncontrolled diabetes and other co morbidities. Motor weakness of upper limbs

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — all-female patients who are home makers
Study Population: All female patients aged between 18-55 years with chronic neck pain (pain lasting for more than 3months) who were homemakers were included in the study. All participants reported presence of pain in the preceeding one week. Homemakers are defined as those who stay at home to care for the home or family. That is, a person irrespective of marital status (married, widowed, divorced, unmarried, separated) with or without children who manages a home and does not earn from employment from either a formal or informal sector.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | 5 minutes
  Visual analogue scale (VAS) is a valid, efficient and convenient measurement tool where subject was asked to mark his or her pain intensity in a 10 cm line divided in gaps of one cm. One end of the line represented no pain while the other signified the' maximum pain experienced by the subject in lifetime'.

SECONDARY OUTCOMES:
The Medical Outcomes Study Short-Form Health Survey (SF 36) | 15 minutes
  The Medical Outcomes Study Short-Form Health Survey (SF 36)is a widely used generic health-related quality of life (QoL) instrument. It has 36 questions measuring health in eight dimensions (physical functioning,role limitations due to physical health problems, bodily pain ,social functioning, general mental health covering psychological distress and well-being (MH), role limitations due to emotional problems , vitality, energy and fatigue and general health perceptions)
Hospital anxiety and depression scale (HADS) | 5 minutes
  Hospital anxiety and depression scale (HADS) is a 14-item questionnaire which assesses both anxiety and depression (7 items each). The score of each subscale [anxiety or depression] can range from 0 to 21. It is used to assess the emotional status.
Work functioning impairment scale) (WFI) | 5 minutes
  Work functioning impairment scale) (WFI) is a a six-item validated instrument that consists of four metrics: absenteeism, presenteeism, overall work productivity loss and activity impairment. Subject was asked to rate in a scale of 1-10 the amount the problem affected their productivity while working.

CONTACTS AND LOCATIONS:
Overall Officials: MADHUSREE SENGUPTA, DNB, PDF, Principal Investigator — CONSULTANT IN NEUROREHABILITATION AT INSTITUTE OF NEUROSCIENCES, KOLKATA, INDIA
Locations (1):
- Institute of Neurosciences Kolkata, Kolkata, West Bengal, India

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers. If required, the Sponsor-Investigator may be contacted via an email shared on this portal